CLINICAL TRIAL: NCT00701584
Title: The Role of Diet, Complementary Treatment and Lifestyle in Breast Cancer Progression and Survival
Brief Title: The Role of Diet and Lifestyle in Breast Cancer Survival
Acronym: DietCompLyf
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College London Hospitals (Other)
Collaborators: United Kingdom Clinical Research Collaboration (Other)
Responsible Party: Director of Research and Developement, UCL Hospitals NHS Foundation Trust
Other Study IDs: 1456
Record Dates: First submitted 2008-06-13; First posted 2008-06-19 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: Phytoestrogens; Isoflavones; Lignans; Breast cancer survival; breast cancer recurrence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, buffy coat, urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Diet has been found to influence hormone production and metabolism which in turn could affect the incidence of hormone related cancers. Consumption of soy-containing foods, known to be rich in phytoestrogens, is thought to be one of the chemoprotective factors against breast cancer in Asian populations. Phytoestrogens have a wide range of metabolic effects and may have a role in effecting breast cancer risk. Although there is mounting evidence of the positive influence of phytoestrogens on breast cancer risk, very little research has been carried out in humans as to the effects of phytoestrogens on breast cancer recurrence and survival. The DietCompLyf study aims to explore this effect by carrying out an observational study in 3,000 breast cancer women in the UK. The effects of diet, lifestyle practices and use of complementary treatments will also be investigated. Participants are recruited 9-15 months post-diagnosis and followed up for 5 years. Questionnaires as well as blood and urine samples are collected annually.

DETAILED DESCRIPTION:
Women matching the eligibility criteria are consented at breast cancer follow-up hospital visits. Blood and urine samples are then collected and questionnaires are provided for the participants to take away and return within 4 weeks. The process of sample collection and questionnaire provision is repeated for visit at years 3 and 5.

Year 2 and 4 study visit vary in that questionnaires including a 7 day food diary are sent to participants at home to be filled in 7 days before their scheduled follow-up appointment. At hospital, blood and urine samples are collected as usual.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed invasive primary breast cancer grades I to III.
* age up to and including 75 years old

Exclusion Criteria:

* Previous cancer with the exception of basal cell carcinoma
* Concomitant primary cancer
* Bilateral cancer of the breast
* Psychological problems
* Cognitive impairment
* Poor understanding of English

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer clinics in UK
Sampling Method: Probability Sample
Enrollment: 3390 (Actual)
Dates: Start 2005-01; Primary Completion 2010-08 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To assess the association between phytoestrogens and relapse free survival | Up to 5 years post-diagnosis

SECONDARY OUTCOMES:
To assess the association between phytoestrogens and event free survival | Up to 5 years post-diagnosis
To assess the association between phytoestrogens and recurrence free survival | Up to 5 years post-diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Miriam V Dwek, PhD, Principal Investigator — University of Westminster
Locations (1):
- University of Westminster, London, United Kingdom